CLINICAL TRIAL: NCT00696839
Title: Clinical Trial Of Cognitive-behavioral Therapy To Reduce Antiretroviral Side Effects In HIV Patients
Brief Title: Trial of Cognitive Behavioral Therapy to Reduce Antiretroviral Therapy Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: R. Eric Doerfler, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: #08-17
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections; Adverse Effects
Keywords: Behavior Therapy; Anti-Retroviral Agents; Relaxation; Clinical Nursing Research; Complementary Therapies
MeSH Terms: conditions — HIV Infections | interventions — Cognitive Behavioral Therapy; Relaxation Therapy; Autogenic Training; Imagery, Psychotherapy; Cognitive Restructuring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Usual care (adherence education)
- 2 (Experimental): Usual care and Cognitive Behavioral Therapy sessions
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — 3 sessions of CBT: introduction of CBT, training in relaxation and guided imagery, and troubleshooting/closure. 50 minute sessions with an HIV-experienced treating psychologist in Beck-type CBT. Participants will be given an audiorecording of the 2nd session to be used in private home practice, as desired.
  Other Names: Relaxation techniques; Progressive muscle relaxation; Guided imagery; Reframing
  Arms: 2

SUMMARY:
The hypothesis is that participants in the intervention group will experience fewer/less intense side effects from anti-HIV medications, if they receive training sessions on the use of guided imagery, relaxation, and reframing of the medication-taking experience. Such training is not part of the usual care of HIV patients.

DETAILED DESCRIPTION:
HIV patients on antiretroviral medications, who are suffering from pain, nausea, anxiety, or fatigue will be randomly assigned to either the usual care for an HIV patient, which is an educational program about the medications, or an intervention program, which includes both the educational program and three sessions with a psychologist. The sessions will help participants understand their concerns about the medications and will teach relaxation techniques and guided imagery to help participants reduce discomforts associated with the medications. All patients will continue to receive the usual care from their medical providers. The main measures are the measured frequency and intensity of the symptoms under study; secondary measures examine medication adherence, CD4 counts, and virus levels. Control measures include the number of doses of side effect medications taken in each group, and the number of relaxation/imagery sessions practiced privately by participants in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Participants currently taking antiretroviral medications for HIV
* Participants suffer from one or more: nausea, pain, fatigue, anxiety

Exclusion Criteria:

* Non-English speaking/reading
* Pregnant or planning to become pregnant within 3 months
* Any severe health problem that would prevent participation (e.g., opportunistic infection requiring hospitalization)
* Substance abuse preventing active participation in care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Side effect symptoms measured by visual analogue scales | study start, 30 days, 60 days, 90 days

SECONDARY OUTCOMES:
Health status by SF-36 | study start, 30 days, 60 days, 90 days
Adherence by visual analogue scale | study start, 30 days, 60 days, 90 days
CD4 lymphocyte count | study start, 90 days
Serum HIV level | study start, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Doerfler, PhD(c), Principal Investigator — Duquesne University School of Nursing
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States